Influence of Custom Orthosis Post Carpometacarpal (CMC) Arthroplasty

# NCT050307510

Document date: document created for submission to UToledo IRB. Approval date of IRB 2/21/22.

## THE ELEMENTS OF A RESEARCH PROTOCOL

# Influence of custom orthosis post CMC arthroplasty

# 1. Background, Review of the Literature, Significance

Carpometacarpal (CMC) osteoarthritis (OA) can cause severe pain and loss of hand function, thumb motion and thumb strength (Fontana et al., 2007). CMC arthroplasty, surgery on the thumb joint, is conducted when conservative treatments for CMC OA fail (Grenier et al. 2016). In 2011, 6,960 CMC arthroplasties were conducted in the United States (Werner et al., 2015). Splints or orthoses are typically used after surgery to immobilize the joint as the wound heals. Previous studies have reported mixed results in the comparison of outcomes related to use of custom orthoses and prefabricated splints (Baradaran et al., 2018; Sillem et al., 2011; Marotta et al., 2020; Bani et al., 2013). This study aims to compare post-surgical outcomes, including wound dehiscence, pain, function, and satisfaction with device and care from individuals who receive either a custom orthosis or prefabricated splint after CMC arthroplasty. This study will allow for increased understanding about the pros and cons of prefabricated splints versus custom orthosis which can inform clinical decisions in order to decrease wound dehiscence, the pain associated with wound dehiscence, and enhance function post-surgery for individuals who have CMC arthroplasty.

# 2. Objectives/Specific Aims

- To determine the difference in the incidence of wound dehiscence after a CMC arthroplasty when using a custom orthosis as compared to a prefabricated splint.
- To determine the difference in subject reported pain levels after a CMC arthroplasty between those who received a custom orthosis as compared to those who received a prefabricated splint.
- To determine the difference in function as measured by the QuickDASH, active range of motion measurements of the thumb, and subtests within the applied dexterity section of the Arthritis Hand Function Test (AHFT) between those wearing a custom orthosis as compared to those wearing a prefabricated splint.
- To determine the difference in subject satisfaction with device and services at the first and second post-operative appointment.

## 3. Methods

# a) Study Design

• Experimental, two groups with random assignment

## b) Method of treatment assignment

Subjects will be randomly assigned using at the initial follow-up appointment following CMC arthroplasty. The surgeon may exclude the subject, following assessment, if the subject cannot be randomly assigned to an intervention group. Open-label blinding will be used since every member of the team will be able to perceive whether the subject has

received a custom orthosis or prefabricated splint. Random assignment to the two groups will be completed in SPSS.

### c) Inclusion/exclusion criteria

Inclusion criteria for subjects include status post CMC arthroplasty (within 4-5 weeks), 18 or older, able to read and understand English, capable of independently consenting to health care procedures.

Subjects will be excluded from the study if the surgeon identifies risk factors that would preclude random assignment to the control or experimental group. Subjects will also be excluded if they request a prefabricated or custom orthosis.

# d) Justification of the number of subjects

Anticipated number of subjects that will be requested for enrollment is 125 subjects. A sample size of at least 96 is required for a power of 60 with  $\alpha = .05$ .

# e) Study setting

University of Toledo Medical Center (UTMC) outpatient.

# f) Primary and secondary outcome measures

Primary Outcomes include:

Function - as measured by the QuickDASH

Wound dehiscence – as measured by the Sandy Grading System

Pain - as measured by the Visual Analog Pain Scale

Thumb CMC Active Range of Motion (AROM) measurements

Subtests within the applied dexterity section of the Arthritis Hand Function Test Satisfaction with device and services – as measured by the OPUS.

Secondary variables of interest include:

Demographic data such as age, gender, race, handedness, pre-existing conditions current medications and supplements, smoking history, and alcohol consumption.

#### h) Procedures, interventions, schedule

#### FIRST POST-OP APPOINTMENT

Standard of care: At the initial post-op appointment with the surgeon, the client will check in and register for the appointment. A member of the surgical team will assess the client and document the Sandy Score.

Research specific: As a member of the surgical team assesses the client he/she will determine if the client meets the inclusion criteria. If the client does meet the inclusion criteria, the study will be briefly explained using the recruitment flyer. The client will then be asked if he/she is interested in participating.

If the client is interested in participating, a member of research team will meet with the client to review the consent form and answer any questions. Once any questions have been answered, if the subject agrees to participate, he/she will sign the informed consent form. The subjects will be informed both verbally and in writing that they can take consent away at any

time during the research study. A copy of the informed consent form will be given to the subject. The client will be randomly assigned to intervention A or intervention B.

Standard of Care: The subject will receive either a prefabricated splint (Intervention A) or custom orthosis (Intervention B).

Research specific: The subject will then be asked to complete the demographic questionnaire, QuickDASH, and the Pain VAS. Thumb CMC active range of motion measurements will then be collected (radial and palmar abduction). Participants will also complete subtests within the applied dexterity section of the Arthritis Hand Function Test and OPUS survey.

Subjects who are assigned to Intervention A (the prefabricated splint group) will be provided a splint by a member of the surgical team. Subjects who are assigned to Invention B (the custom orthosis group) will be evaluated by an occupational therapist and a custom orthosis will be fabricated.

#### SECOND POST-OP APPOINTMENT

Standard of Care: Approximately 4-5 weeks later, subjects will attend a second post-op appointment and be assessed by a member of the surgical team. The Sandy score will be documented.

Research specific: At this time, a member of the research team will ask the subject to complete the, QuickDASH, and the Pain VAS. Thumb CMC active range of motion measurements will then be collected (radial and palmar abduction). Participants will also complete subtests within the applied dexterity section of the Arthritis Hand Function Test and OPUS survey.

## i) Planned data analysis

Means and standard deviations will be calculated for the demographic information such as age and alcohol consumption per week. In-group and between-group percentages will also be calculated for demographic information, such as gender, pre-existing diabetes, and smoking history. The means and standard deviations of scores received on the QuickDASH, Sandy Grading System, Pain VAS, and AROM will be calculated. In-group and between-group descriptive statistics will be calculated for scores on the OPUS and Applied Dexterity section of the Arthritis Hand Function test. Independent student t-tests will be conducted to compare the means between Interventions A and B. Dependent student t-tests will be conducted to compare the initial post-op assessment mean data to the second post-op assessment mean data within groups. P-values will be considered significant if they are less than or equal to 0.05.

#### 4. Reference List

Aebischer, B., Elsig, S., & Taeymans, J. (2016). Effectiveness of physical and occupational therapy on pain, function and quality of life in patients with trapeziometacarpal osteoarthritis - A systematic review and meta-analysis. *Hand therapy*, 21(1), 5–15. <a href="https://doi.org/10.1177/1758998315614037">https://doi.org/10.1177/1758998315614037</a>

Baca, M. E., Rozental, T. D., McFarlane, K., Hall, M. J., Ostergaard, P. J., & Harper, C. M. (2020). Trapeziometacarpal joint arthritis: is duration of symptoms a predictor of

- surgical outcomes? *The Journal of Hand Surgery, 45*(12), 1184.e1-1184.e7. https://doi.org/10.1016/j.jhsa.2020.05.026
- Bani, M. A., Arazpour, M., Kashani, R. V., Mousavi, M. E., & Hutchins, S. W. (2013). Comparison of custom-made and prefabricated neoprene splinting in patients with the first carpometacarpal joint osteoarthritis. *Disability & Rehabilitation: Assistive Technology*, 8(3), 232–237. <a href="https://doi.org/10.3109/17483107.2012.699992">https://doi.org/10.3109/17483107.2012.699992</a>
- Bani, M. A., Arazpour, M., Kashani, R. V., Mousavi, M. E., Maleki, M., & Hutchins, S. W. (2013). The effect of custom-made splints in patients with the first carpometacarpal joint osteoarthritis. *Prosthetics and Orthotics International*, *37*(2), 139–144. <a href="https://doi.org/10.1177/0309364612454047">https://doi.org/10.1177/0309364612454047</a>
- Baradaran, A., Baradaran, A., Ebrahimzadeh, M. H., Kachooei, A. R., Rivlin, M., & Beredjiklian, P. (2018). Comparison of custom-made versus prefabricated thumb splinting for carpometacarpal arthrosis: A systematic review and meta-analysis. *The Archives Of Bone And Joint Surgery*, 6(6), 478–485.
- Barnard, A. R., Regan, M., Burke, F. D., Chung, K. C., & Wilgis, E. F. S. (2012). Wound healing with medications for rheumatoid arthritis in hand surgery. *ISRN Rheumatology*, 2012, 251962. https://doi.org/10.5402/2012/251962.
- Becker, S. J., Bot, A. G., Curley, S. E., Jupiter, J. B., & Ring, D. (2013). A prospective randomized comparison of neoprene vs thermoplast hand-based thumb spica splinting for trapeziometacarpal arthrosis. *Osteoarthritis and cartilage*, 21(5), 668–675. <a href="https://doi.org/10.1016/j.joca.2013.02.006">https://doi.org/10.1016/j.joca.2013.02.006</a>
- Berggren, M., Joost-Davidsson, A., Lindstrand, J., Nylander, G., & Povlsen, B. (2001).

  Reduction in the need for operation after conservative treatment of osteoarthritis of the first carpometacarpal joint: A seven year prospective study. *Scandinavian journal of plastic and reconstructive surgery and hand surgery*, 35(4), 415–417. <a href="https://doi.org/10.1080/028443101317149381">https://doi.org/10.1080/028443101317149381</a>
- Bertozzi, L., Valdes, K., Vanti, C., Negrini, S., Pillastrini, P., & Villafañe, J. H. (2015). Investigation of the effect of conservative interventions in thumb carpometacarpal osteoarthritis: Systematic review and meta-analysis. *Disability and Rehabilitation*, 37(22), 2025–2043. https://doi.org/10.3109/09638288.2014.996299
- Boonstra, A. M., Schiphorst Preuper, H. R., Reneman, M. F., Posthumus, J. B., & Stewart, R. E. (2008). Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. *International journal of rehabilitation research*. *Internationale Zeitschrift fur Rehabilitationsforschung*. *Revue internationale de recherches de readaptation*, 31(2), 165–169. <a href="https://doi.org/10.1097/MRR.0b013e3282fc0f93">https://doi.org/10.1097/MRR.0b013e3282fc0f93</a>
- Crosby, C. A., Reitz, J. L., Mester, E. A., & Grenier, M.-L. (2013). Rehabilitation following thumb CMC, radiocarpal, and DRUJ arthroplasty. *Hand Clinics*, *29*(1), 123–142. <a href="https://doi.org/10.1016/j.hcl.2012.08.025">https://doi.org/10.1016/j.hcl.2012.08.025</a>
- Day, C. S., Gelberman, R., Patel, A. A., Vogt, M. T., Ditsios, K., & Boyer, M. I. (2004). Basal joint osteoarthritis of the thumb: a prospective trial of steroid injection and splinting. *The Journal of Hand Surgery*, 29(2), 247–251. https://doi.org/10.1016/j.jhsa.2003.12.002
- De Smet, L., Sioen, W., Spaepen, D., & van Ransbeeck, H. (2004). Treatment of basal joint arthritis of the thumb: Trapeziectomy with or without tendon interposition/ligament reconstruction. *Hand Surgery*, 9(1), 5–9. <a href="https://doi.org/10.1142/S0218810404001942">https://doi.org/10.1142/S0218810404001942</a>
- Earp, B. E. (2008). Treatment of advanced CMC joint disease: Trapeziectomy and implant arthroplasty (silastic-metal-synthetic allograft). *Hand Clinics*, 24(3), 277. <a href="https://doi.org/10.1016/j.hcl.2008.04.004">https://doi.org/10.1016/j.hcl.2008.04.004</a>

- Field, J., Buchanan, D. (2007). To suspend or not to suspend: a randomised single blind trial of simple trapeziectomy versus trapeziectomy and flexor carpi radialis suspension. *J Hand Surg Eur* 32(4), 462-466. doi.10.1016/J.JHSB.2007.02.005
- Fontana, L., Neel, S., Claise, J.-M., Ughetto, S., & Catilina, P. (2007). Osteoarthritis of the thumb carpometacarpal joint in women and occupational risk factors: A case-control study. *The Journal of Hand Surgery*, 32(4), 459–465. <a href="https://doi.org/10.1016/j.jhsa.2007.01.014">https://doi.org/10.1016/j.jhsa.2007.01.014</a>
- Frye, S. K., & Geigle, P. R. (2020). A comparison of prefabricated and custom made resting hand splints for individuals with cervical spinal cord injury: A randomized controlled trial. *Clinical rehabilitation*, 269215520983486. Advance online publication. https://doi.org/10.1177/0269215520983486
- Grenier, M. L., Mendonca, R., & Dalley, P. (2016). The effectiveness of orthoses in the conservative management of thumb CMC joint osteoarthritis: An analysis of functional pinch strength. *Journal of hand therapy: official journal of the American Society of Hand Therapists*, 29(3), 307–313. https://doi.org/10.1016/j.jht.2016.02.004
- Gummesson, C., Ward, M. M., & Atroshi, I. (2006). The shortened disabilities of the arm, shoulder and hand questionnaire (QuickDASH): Validity and reliability based on responses within the full-length DASH. *BMC musculoskeletal disorders*, 7, 44. https://doi.org/10.1186/1471-2474-7-44
- Halilaj, E., Moore, D. C., Laidlaw, D. H., Got, C. J., Weiss, A.-P. C., Ladd, A. L., & Crisco, J. J. (2014). The morphology of the thumb carpometacarpal joint does not differ between men and women, but changes with aging and early osteoarthritis. *Journal of Biomechanics*, 47(11), 2709–2714. https://doi.org/10.1016/j.jbiomech.2014.05.005
- Hamann, N., Heidemann, J., Heinrich, K., Wu, H., Bleuel, J., Gonska, C., & Brüggemann, G.
  P. (2014). Stabilization effectiveness and functionality of different thumb orthoses in female patients with first carpometacarpal joint osteoarthritis. *Clinical biomechanics* (*Bristol, Avon*), 29(10), 1170–1176. <a href="https://doi.org/10.1016/j.clinbiomech.2014.09.007">https://doi.org/10.1016/j.clinbiomech.2014.09.007</a>
- Kooner, S. S., Sheehan, B., Kendal, J. K., & Johal, H. (2018). Development of a simple multidisciplinary arthroplasty wound-assessment instrument: the SMArt Wound Tool. Canadian Journal of Surgery. Journal Canadian de Chirurgie, 61(5), 326–331. <a href="https://doi.org/10.1503/cjs.015017">https://doi.org/10.1503/cjs.015017</a>
- London, D. A., Stepan, J. G., Lalchandani, G. R., Okoroafor, U. C., Wildes, T. S., & Calfee, R. P. (2014). The impact of obesity on complications of elbow, forearm, and hand surgeries. *The Journal of Hand Surgery*, *39*(8), 1578–1584. https://doi.org/10.1016/j.jhsa.2014.05.007
- Marotta, N., Demeco, A., Marinaro, C., Moggio, L., Pino, I., Barletta, M., Petraroli, A., & Ammendolia, A. (2020). Comparative effectiveness of orthoses for thumb osteoarthritis: A systematic review and network meta-analysis. *Archives of Physical Medicine and Rehabilitation*. https://doi.org/10.1016/j.apmr.2020.06.012
- Matullo, K. S., Ilyas, A., & Thoder, J. J. (2007). CMC arthroplasty of the thumb: A review. *Hand* (New York, N.Y.), *2*(4), 232–239. <a href="https://doi.org/10.1007/s11552-007-9068-9">https://doi.org/10.1007/s11552-007-9068-9</a>
- McKee, P., & Rivard, A. (2004). Orthoses as enablers of occupation: client-centred splinting for better outcomes. *Canadian Journal of Occupational Therapy*, 71(5), 306–314.
- Ooishi, D., Izumi, M., Ueba, H., & Ikeuchi, M. (2019). Splinting for the carpometacarpal joint relieves experimental basal thumb pain and loss of pinch strength. *European Journal of Pain (London, England)*, 23(7), 1351–1357. https://doi.org/10.1002/ejp.1404
- Poole, J. L., Walenta, M. H., Alonzo, V., Coe, A., & Moneim, M. (2011). A pilot study comparing of two therapy regimens following carpometacarpal joint

- arthroplasty. *Physical & Occupational Therapy in Geriatrics*, 29(4), 327–336. https://doi.org/10.3109/02703181.2011.613530
- Rannou, F., Dimet, J., Boutron, I., Baron, G., Fayad, F., Macé, Y., Beaudreuil, J., Richette, P., Ravaud, P., Revel, M., & Poiraudeau, S. (2009). Splint for base-of-thumb osteoarthritis: A randomized trial. *Annals of Internal Medicine*, *150*(10), 661–669.
- Rhee, P. C., Paul, A., Carlsen, B., & Shin, A. Y. (2019). Outcomes of surgical management for thumb basilar arthritis in patients 55 years of age and younger. *Hand* (New York, N.Y.), *14*(5), 641–645. https://doi.org/10.1177/1558944718769378
- Roberts, R. A., Jabaley, M. E., & Nick, T. G. (2001). Results following trapeziometacarpal arthroplasty of the thumb. *Journal of Hand Therapy: Official Journal of the American Society of Hand Therapists*, 14(3), 202–207. https://doi.org/10.1016/s0894-1130(01)80054-5
- Rosen, R., Manna, B. (2020). Wound Dehiscence. *StatPearls Publishing*. <a href="https://www.ncbi.nlm.nih.gov/books/NBK551712/">https://www.ncbi.nlm.nih.gov/books/NBK551712/</a>
- Sandy-Hodgetts, K., Carville, K., Santamaria, N., Parsons, R., & Leslie, G. D. (2019). The Perth Surgical Wound Dehiscence Risk Assessment Tool (PSWDRAT): Development and prospective validation in the clinical setting. *Journal of Wound Care*, 28(6), 332–344. <a href="https://doi.org/10.12968/jowc.2019.28.6.332">https://doi.org/10.12968/jowc.2019.28.6.332</a>
- Sandy-Hodgetts, K., Ousey, K., Conway, B., Djohan, R., Nair, H. K. R., Serena, T. E., & Tariq, G. (2020). International best practice recommendations for the early identification and prevention of surgical wound complications. London, UK; Wounds International. <a href="https://iswcap.org/wp-content/uploads/2020/03/ESS20">https://iswcap.org/wp-content/uploads/2020/03/ESS20</a> CD ISWCAP WINT web.pdf
- Shah, K. N., Defroda, S. F., Wang, B., & Weiss, A.-P. C. (2019). Risk factors for 30-day complications after thumb CMC joint arthroplasty: An American College of Surgeons national surgery quality improvement program study. *Hand*, *14*(3), 357–363. <a href="https://doi.org/10.1177/1558944717744341">https://doi.org/10.1177/1558944717744341</a>
- Siegel, P., Jackson, D., & Baugh, C. (2020). Practice patterns following carpometacarpal (CMC) arthroplasty. *Journal of hand therapy: official journal of the American Society of Hand Therapists*, S0894-1130(20)30206-4. Advance online publication. <a href="https://doi.org/10.1016/j.jht.2020.10.016">https://doi.org/10.1016/j.jht.2020.10.016</a>
- Sillem, H., Backman, C. L., Miller, W. C., & Li, L. C. (2011). Comparison of two carpometacarpal stabilizing splints for individuals with thumb osteoarthritis. *Journal of hand therapy: Official journal of the American Society of Hand Therapists*, 24(3), 216–230. <a href="https://doi.org/10.1016/j.jht.2010.12.004">https://doi.org/10.1016/j.jht.2010.12.004</a>
- Silva, P. G., De Carvalho Silva, F., Da Rocha Corrêa Fernandes, A., & Natour, J. (2020). Effectiveness of nighttime orthoses in controlling pain for women with hand osteoarthritis: A randomized controlled trial. *American Journal of Occupational Therapy*, 74(3), 7403205080p1. <a href="https://doi.org/10.5014/ajot.2020.033621">https://doi.org/10.5014/ajot.2020.033621</a>
- Thomsen, N. O., Jensen, C. H., & Nygaard, H. (2000). Weilby-Burton arthroplasty of the trapeziometacarpal joint of the thumb. *Scandinavian Journal of Plastic and Reconstructive Surgery and Hand Surgery*, 34(3), 253–256. https://doi.org/10.1080/02844310050159846
- Tsehaie, J., Wouters, R. M., Feitz, R., Slijper, H. P., Hovius, S. E. R., & Selles, R. W. (2019). Shorter vs longer immobilization after surgery for thumb carpometacarpal osteoarthritis: A propensity score-matched study. *Archives of Physical Medicine and Rehabilitation*, 100(11), 2022. https://doi.org/10.1016/j.apmr.2019.02.016
- Vermeulen, G. M., Brink, S. M., Sluiter, J., Elias, S. G., Hovius, S. E. R., & Moojen, T. M. (2009). Ligament reconstruction arthroplasty for primary thumb carpometacarpal

- osteoarthritis (Weilby technique): Prospective cohort study. *Journal of Hand Surgery*, 34(8), 1393–1401. https://doi.org/10.1016/j.jhsa.2009.06.019
- Weiss, S., Lastayo, P., Mills, A., & Bramlet, D. (2004). Splinting the degenerative basal joint: Custom-made or prefabricated neoprene? *Journal of Hand Therapy*, 17(4), 401–406. <a href="https://doi.org/10.1197/j.jht.2004.07.002">https://doi.org/10.1197/j.jht.2004.07.002</a>
- Werner, B. C., Bridgforth, A. B., Gwathmey, F. W., & Dacus, A. R. (2015). Trends in thumb carpometacarpal interposition arthroplasty in the United States, 2005-2011. *American Journal of Orthopedics* (Belle Mead, N.J.), 44(8), 363–368.
- Witherow, E. J., & Peiris, C. L. (2015). Custom-made finger orthoses have fewer skin complications than prefabricated finger orthoses in the management of mallet injury: A systematic review and meta-analysis. *Archives of physical medicine and rehabilitation*, 96(10), 1913–1923.e1. https://doi.org/10.1016/j.apmr.2015.04.026
- Wollstein, R., Michael, D., & Harel, H. (2015). Postoperative therapy for chronic thumb carpometacarpal (CMC) joint dislocation. *American Journal of Occupational Therapy*, 70(1), 7001350020p1. <a href="https://doi.org/10.5014/ajot.2016.017210">https://doi.org/10.5014/ajot.2016.017210</a>
- Youngman, T., Del Core, M., Benage, T., Koehler, D., Sammer, D., & Golden, A. (2020). Patient-related risk factors associated with surgical site complications after elective hand surgery. *Hand* (New York, N.Y.), 1558944720944260. https://doi.org/10.1177/1558944720944260